CLINICAL TRIAL: NCT03741452
Title: Evaluation of Ultrasound-guided Transversalis Fascia Plane Block for Postoperative Analgesia in Cesarean Section: A Prospective, Randomized, Controlled Clinical Trial
Brief Title: Transversalis Fascia Plane Block in Caesarean Section Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maltepe University (Other)
Responsible Party: Principal Investigator, Asst. Prof. Serkan Tulgar, M.D., assoc professor in anesthesiology and reanimation, Maltepe University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TFPB in CS
Record Dates: First submitted 2018-11-11; First posted 2018-11-14 (Actual); Last update posted 2019-02-25 (Actual); Status verified 2018-11

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Analgesia, Patient-Controlled

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transversalis fascia plane block (Experimental): The transversalis fascia plane block will be administrated to this group at end of the surgery under general anesthesia. An intravenous patient-controlled analgesia device within tramadol will be given to the patients postoperatively.
  Interventions: Other: transversalis fascia plane block
- Control group (No Intervention): In this group, patients will receive only multimodal analgesic treatment including patient-controlled analgesia with tramadol. No block will be performed.

INTERVENTIONS:
Other: transversalis fascia plane block — patient controlled analgesia devices with tramadol
  Other Names: patient controlled analgesia
  Arms: Transversalis fascia plane block

SUMMARY:
Transversalis fascia plane block is a regional anesthesia technique described ten years ago. Its use for many indications has been identified by case reports in the literature. As the investigators have considered that transversalis fascia plane block could be efficacious for providing postoperative analgesia in the cesarean section, the investigators have implemented the application of this blockade into practice at the clinic. The main purpose of this study is to evaluate the analgesic effect of ultrasound-guided bilateral transversalis fascia plane block in cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing cesarean section under general anesthesia ASA I-II

Exclusion Criteria:

* patients undergoing cesarean section under neuraxial anesthesia morbidly obesity ASA III - IV infection of the skin at the site of needle puncture area patients with known allergies to any of the study drugs coagulopathy recent use of analgesic drugs

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2018-11-26 (Actual); Primary Completion 2019-02-19 (Actual); Study Completion 2019-02-22 (Actual)

PRIMARY OUTCOMES:
24 hours tramadol consumption | 24 hour
  tramadol consumptions for both group will be recorded

SECONDARY OUTCOMES:
Numeric rating scale for postoperative pain intensity | 24 hours
  Changes in Numeric Rating Scale (NRS) at rest and on movement will be recorded at intervals. NRS is a unidimensional measure of pain intensity in adults. The NRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain. The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").
Postoperative nausea and vomiting | 24 hours
  number of postoperative nasusea and vomiting after surgery will be questioned

CONTACTS AND LOCATIONS:
Locations (1):
- Maltepe University faculty of medicine, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tulgar S, Serifsoy TE. Transversalis fascia plane block provides effective postoperative analgesia for cesarean section: New indication for known block. J Clin Anesth. 2018 Aug;48:13-14. doi: 10.1016/j.jclinane.2018.04.006. Epub 2018 Apr 22. No abstract available. PMID 29689328
- [Background] Sondekoppam RV, Ip V, Johnston DF, Uppal V, Johnson M, Ganapathy S, Tsui BCH. Ultrasound-guided lateral-medial transmuscular quadratus lumborum block for analgesia following anterior iliac crest bone graft harvesting: a clinical and anatomical study. Can J Anaesth. 2018 Feb;65(2):178-187. doi: 10.1007/s12630-017-1021-y. Epub 2017 Nov 21. PMID 29164530